CLINICAL TRIAL: NCT00945503
Title: An Adaptive PET Study in Healthy Volunteers Using [11C]GSK931145 to Establish the Relationship of Glycine Transporter 1 Occupancy by GSK1018921 to Plasma Concentrations Over Time.
Brief Title: Positron Emission Tomography (PET) Study to Describe the Relationship Between Plasma Concentrations and Brain Gly-T1 Occupancy of GSK1018921 Over Time.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109731
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Schizophrenia
Keywords: Glycine Tranporter; MRI; PET
MeSH Terms: conditions — Schizophrenia | interventions — GSK 1018921

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK1018921 (Experimental): All subjects will received a dose of GSK1018921 and will peforme three PET scans using the ligand [11C]GSK931145, but in order to obtain adequate sampling of the exposure-time-occupancy curves, a range of doses will be evaluated, and the timing of the post-dose scans will differ between subjects.
  Interventions: Drug: GSK1018921

INTERVENTIONS:
Drug: GSK1018921 — GSK1018921 is a GT1 recepor antagonist

SUMMARY:
A PET study using [11c]GSK931145 to characterise the exposure-occupancy relationship over time for GSK1018921.

DETAILED DESCRIPTION:
This is an open-label, adaptive-design, single-dose, non randomized PET occupancy study.The primary aim of this study is to describe the relationship between plasma concentrations and brain occupancy of GSK1018921 over time. Up to 22 healthy volunteers will be administered single doses of GSK1018921 in order to obtain 12 evaluable complete data sets of occupancy estimates.

ELIGIBILITY:
* Inclusion criteria:

  * Healthy male subjects
  * Age: 18-55 years
  * No history of physical, neurological or mental illness
* Exclusion criteria

  * History of claustrophobia or inability to lie still in the PET camera for at least 2 hours
  * Cardiac pacemakers or metal implants in the body that contraindicate MRI scan.
  * History of regular alcohol consumption (weekly intake >21 units) within the previous six months.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-05-19 (Actual); Primary Completion 2008-12-22 (Actual); Study Completion 2008-12-22 (Actual)

PRIMARY OUTCOMES:
PET occupancy with GSK1018921 | 10 days

SECONDARY OUTCOMES:
To assess the safety the AEs and SAEs will be collected during the study such as vital signs, physical exams and laboratory safety tests. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 109731 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/109731?search=study&search_terms=109731#rs
- Available data/document: Annotated Case Report Form: 109731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register